CLINICAL TRIAL: NCT04481425
Title: Evaluation of the Efficacy of Non-drug Therapy (SMS Intervention) for Adolescents With NSSI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Jian-Jun Ou, Principal Investigator, Central South University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MD20200309
Record Dates: First submitted 2020-07-13; First posted 2020-07-22 (Actual); Last update posted 2022-11-18 (Actual); Status verified 2022-11

CONDITIONS: Non-suicidal Self-injury
MeSH Terms: conditions — Self-Injurious Behavior

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Other): Text messages will be sent to the subjects through the investigator, including giving popularization of psychiatric knowledge, coping skills, emotional regulation strategies, and brief care. Two or three times a week for two months.
  Interventions: Other: SMS intervention
- control group (No Intervention): Subjects both collected in the outpatient department and the ward were randomly divided into the control group and regularly followed up.

INTERVENTIONS:
Other: SMS intervention — SMS intervention
  Arms: intervention group

SUMMARY:
In this proposed study, Text messages are used to intervene in the NSSI behavior of adolescents, and the efficacy of this intervention method is evaluated, as well as the internal mechanism of adolescents' NSSI behavior is discussed.

DETAILED DESCRIPTION:
In this proposed study, the investigators will evaluate the effect of text message intervention on Nonsuicidal self-injury behavior in adolescents. The study will recruit 110 adolescents with Nonsuicidal self-injury behavior in outpatient and ward, then all the participants will be randomized to the intervention group (55 cases) or the control group 55 cases) for an 8-week clinic trial. Clinical efficacy and safety assessment will be done at baseline, the fourth week, and the eighth week. The specific aims are to evaluate the effect of text message intervention on NSSI in adolescents are on 1) Tendency and frequency of Nonsuicidal self-injury behavior; 2) Level of negative emotion such as depression, anxiety, and hopelessness 3) The use of emotion regulation strategies and coping styles. A semi-structured quantitative interview will be conducted among adolescents from the SMS group to get the attitude and experiences feedback about the text message.

ELIGIBILITY:
Inclusion Criteria:

1. Adolescents aged 10-19 years old.
2. Meet the diagnostic criteria of NSSI behavior recommended by DSM-5.
3. The adolescents who have mobile phone, and have the ability to send or receive text messages.
4. Adolescents and guardians agreed to participate and signed the informed consent form

Exclusion Criteria:

1. Adolescents with severe somatic diseases who cannot complete the study.
2. Adolescents with cognitive impairment, neurodevelopmental disorder, mental retardation, visual impairment who cannot complete the study.
3. The adolescents who do not have a mobile phone.

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 86 (Actual)
Dates: Start 2020-12-23 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
The change of NSSI behavior of the participants. | At baseline, the fourth week, the eighth week
  NSSI behavior will be measured by Nonsuicidal self-injury Questionnaire which contains several items designed by investigators. The questionnaire is mainly used to measure the frequency of NSSI among adolescents.

SECONDARY OUTCOMES:
The change of anxiety level. | At baseline, the fourth week, the eighth week
  The Generalized Anxiety Disorder 7-item Scale will be used to measure the change of anxiety. GAD-7 scale consists of 7 items. Each item ranging from 0 to 3, and the total score ranging from 0 to 21. The higher score indicates severe anxiety symptoms.
The change of depression level. | At baseline, the fourth week, the eighth week
  The Patient Health Questionnaire 9-item will be used to measure the change of depression. PHQ-9 scale consists of 9 items. Each item raging from 0 to 3, and the total score ranging from 0 to 27. The higher score indicates severe depression symptoms.
The change of hopelessness. | At baseline, the fourth week, the eighth week
  The Beck Hopelessness Scale will be used to measure the change of hopelessness. BHS scale consists of 20 items. Each item can be answered "yes" or "no" for 1 or 0 points respectively. The total score ranging from 0 to 20. A higher total score indicates a higher degree of hopelessness.
The change of emotion regulation strategies. | At baseline, the fourth week, the eighth week
  The Emotion Regulation Questionnaire will be used to measure the change of emotion regulation styles. ERQ scale consists of 10 items which can be divided into cognitive reappraisal and expression suppression two emotion-regulating strategy subscales. Each item ranging from 1 to 7 points. The higher the score, the more often the respondent used this emotion-regulating strategy.
The change of coping styles. | At baseline, the fourth week, the eighth week
  The Simplified Coping Style Questionnaire will be used to measure the change of coping styles. SCSQ scale consists of 20 items which can be divide into positive coping styles and negative coping styles in two dimensions. Each item raging from 0 to 3, and the total score ranging from 0 to 60. The higher the score, the more likely the respondents are to use this coping style.
The change of life events stress. | At baseline, the fourth week, the eighth week
  The Adolescent Self-Rating Life Events Check-list will be used to measure the frequency and intensity of life events that may trigger a stressful psychological response in adolescents. There are 27 items in the scale, which can be divided into 6 dimensions. The scale scores ranged from 27 to 135. The higher the score means the higher the degree of negative life event stress. The scale is widely used in China and has good reliability and validity.

CONTACTS AND LOCATIONS:
Overall Officials: Jianjun Ou, doctor, Study Chair — Central South University; Runsen Chen, doctor, Study Director — Central South University
Locations (1):
- Department of Psychiatry, Xiangya Second Hospital, Central South University, Changsha, Hunan, China